CLINICAL TRIAL: NCT02800980
Title: Management of Symptomatic Post-operative Lymphocele With an Patient-controlled, Vascular Catheter: A Validation Study
Brief Title: Management of Symptomatic Post-operative Lymphocele
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maciej Stukan, MD, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Maciej Stukan, MD, PhD, Dr, Gdynia Oncology Center
Organization: Gdynia Oncology Center (Other Government)
Other Study IDs: GCO-3
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Lymphocele
Keywords: lymphocele; sclerotherapy; drainage; percutaneous
MeSH Terms: conditions — Lymphocele | interventions — Drainage; Sclerotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Drainage and sclerotherapy.: Patients with symptomatic lymphocele who are managed with percutaneous drainage and sclerotherapy.
  Interventions: Procedure: Drainage and sclerotherapy.
- Drainage alone.: Patients with symptomatic lymphocele who are managed with percutaneous drainage alone.
  Interventions: Procedure: Drainage alone.

INTERVENTIONS:
Procedure: Drainage and sclerotherapy. — Lymphocele percutaneous / transvaginal drainage with a use of a vascular catheter followed by sclerotherapy.
  Groups: Drainage and sclerotherapy.
Procedure: Drainage alone. — Lymphocele percutaneous / transvaginal drainage with a vascular catheter alone (without sclerotherapy).
  Groups: Drainage alone.

SUMMARY:
Symptomatic lymphocele (LC) can be a complication after pelvic and para-aortic lymphadenectomy performed for treatment or staging purposes in the management of some cancers. Management procedures are: single or repeated puncture, prolonged drainage with drains or catheters, mostly followed by sclerotherapy, or surgery. A decision, which management option is most optimal, should be guided by two principles: first to control patient's symptoms, second to apply the least invasive but effective way to treat LC, taking into account that the patient has undergone major surgery recently, and often needs adjuvant treatment at the moment when symptomatic LC is diagnosed.

The aim of this study is to validate feasibility, safety and efficacy of a minimally invasive management of a symptomatic LC - drainage with the usage of vascular catheter followed by sclerotherapy, as well as to evaluate patient's experience on the treatment.

Patients with symptomatic LC are evaluated with ultrasound. Data about diameters, estimated volume of LC and other organs failure if appear is recorded. Management options are discussed with patient, and if the method with catheter insertion and drainage is chosen than the patient is eligible for the study. After vascular catheter insertion into LC and fluid evacuation, patient is followed with active drainage. Patients with drainage only are observed for a short period of time (up to 7 days), and if not efficient a sclerotherapy is considered. In case a patient does not agree to sclerotherapy, or there are contraindications, or it is doctor's decision that drainage alone is sufficient, than the prolonged drainage without sclerotherapy is the only procedure. The choice about the regimen used for sclerotherapy, it's volume, time intervals between repeated infusion depend on institution practice.

Data concerning feasibility, safety and efficacy are noted in designated templates. Patients' experience on the treatment is evaluated with formal questionnaire FACIT-TS-G.

The study is observational. Primary outcome measure is to establish efficacy of the method. Secondary outcome measures are safety and patient's experience on the treatment.

Investigators hope to establish step-by-step guidelines for optimal, minimally invasive management of symptomatic lymphocele.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic lymphocele after abdominal lymphadenectomy for cancer,
* age > 18 years old,
* informed consent signed,

Exclusion Criteria:

* asymptomatic lymphocele,
* apparent infection of the skin or subcutaneus tissue over the lymphocele (in the place of potential catheter insertion),
* significant coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a symptomatic lymphocele after retroperitoneal, abdominal, pelvic lymphadenectomy for treatment or staging procedures for cancer management.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful lymphocele treatment. | 2 months
  Successful lymphocele treatment means complete resolution of lymphocele after minimally invasive procedures - percutaneous drainage with a vascular catheter followed by sclerotherapy or drainage alone. Opposite - non successful treatment defined when the patient is refered for a surgical management.

SECONDARY OUTCOMES:
Number of successful catheter insertion into lymphocele lumen. | 1 day
Number of adverse events concerned with catheter insertion. | 2 months
Number of adverse events concerned with sclerotherapy. | 2 months

OTHER OUTCOMES:
Patient's experience on the treatment. | 2 months.
  measured with a questionnaire FACIT-TS-G (Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General) available from http://www.facit.org/facitorg/questionnaires. Permission to use obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Stukan, Principal Investigator — Gdynia Oncology Center
Locations (1):
- Gdynia Oncology Center, Gdynia, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stukan M, Dudziak M. Lymphocele in gynecologic oncology practice - management and prophylaxis. Nowotwory Journal of Oncology 61 (3): 272-278, 2011.
- [Result] Mahrer A, Ramchandani P, Trerotola SO, Shlansky-Goldberg RD, Itkin M. Sclerotherapy in the management of postoperative lymphocele. J Vasc Interv Radiol. 2010 Jul;21(7):1050-3. doi: 10.1016/j.jvir.2010.03.014. Epub 2010 Jun 2. PMID 20537556
- [Result] Stukan M, Lesniewski-Kmak K, Wroblewska M, Dudziak M. Management of symptomatic ascites and post-operative lymphocysts with an easy-to-use, patient-controlled, vascular catheter. Gynecol Oncol. 2015 Mar;136(3):466-71. doi: 10.1016/j.ygyno.2014.11.073. Epub 2014 Nov 28. PMID 25434633
- See also: A video step-by-step procedure of vascular catheter insertion into lymphocele lumen followed by sclerotherapy. — https://medtube.net/gynecology/medical-videos/16554-